CLINICAL TRIAL: NCT06706557
Title: A Pilot Study on the Analysis of Circulating Tumor DNA (ctDNA) in HER2-low Advanced/Metastatic Breast Cancer
Brief Title: Analysis of Circulating Tumor DNA (ctDNA) in HER2-low Advanced/Metastatic Breast Cancer
Acronym: LEGO
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1990
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Advanced Metastatic Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Pilot study on circulating tumor DNA (ctDNA) in advanced/metastatic breast cancer with low levels of HER2 expression (HER2 low)

DETAILED DESCRIPTION:
Prospective single-center feasibility study of 30 patients with carcinoma breast with low levels of HER2 expression, defined as 1+ or 2+ expression levels by the IHC technique (immunohistochemistry) and the gene not amplified by the ISH test (in situ hybridization)

ELIGIBILITY:
Inclusion Criteria

* Participants diagnosed with HER2-low breast cancer, defined as IHC score 1+ or 2+ and not amplified at in situ hybridization (ISH) test as confirmed by local laboratory testing.
* Participants should be at advanced or metastatic setting prior to treatment.
* Written informed consent (Accordo di Partecipazione alla Ricerca Scientifica) and specific informed consent to the study must be signed and dated by the patient and the doctor prior to inclusion.
* Patients must be accessible for follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced/metastatic breast cancer with low levels of HER2 expression (HER2 low)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
circulating tumor DNA (ctDNA) in advanced/metastatic breast cancer with low levels of HER2 expression (HER2 low) | 12 months
  evaluate the mutations present in breast cancer of patients with advanced/metastatic disease e HER2-low defined with 1+ or 2+ expression levels by IHC (immunohistochemistry) technique and gene not amplified by ISH test (in situ hybridization)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fusco, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, MI, Italy